CLINICAL TRIAL: NCT03327545
Title: Clinical Efficacy of Mobilization of the Nervous System Compared to Soft Tissue Techniques Intervention in Asymptomatic Subjects With Latent Myofascial Trigger Points in the Craniocervical Region: a Randomized Controlled Trial
Brief Title: Latent Myofascial Trigger Points in the Craniocervical Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LMTrP
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Myofascial Pain Syndrome
Keywords: Trigger points; Trigegeminal nerve; Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): Neural mobilization for a total of 12 minutes
  Interventions: Device: Neural mobilization
- Experimental Group 2 (Experimental): Soft tissue techniques and Stretching right side of the craniocervical for a total of 12 minutes
  Interventions: Device: Soft tissue techniques and Stretching
- Control group (Placebo Comparator): Control group
  Interventions: Device: Control group

INTERVENTIONS:
Device: Neural mobilization — Neural mobilization on the right side of the craniocervical region for a total of 12 minutes.
  Arms: Experimental Group 1
Device: Soft tissue techniques and Stretching — Soft tissue techniques and Stretching on the right side of the craniocervical region for a total of 12 minutes
  Arms: Experimental Group 2
Device: Control group — Did not receive any treatment.
  Arms: Control group

SUMMARY:
Myofascial pain is a clinical problem that has generated interest, debate and confusion for decades. According to studies anywhere between 33 and 97 % of patients with musculoskeletal pain visiting physicians and manual therapists are diagnosed with Myofascial Trigger Points (MTrPs). MTrPs are localized, hyperirritable points that are associated with palpable nodules in taut bands (TB) of muscle fibres. MTrPs can be classified into active and latent. Latent MTrPs demonstrate the same clinical characteristics as active MTrPs but they do not provoke spontaneous pain. The myofascial trigger points (MTrPs) are common in healthy subjects and in patients with musculoskeletal pain, and could produce sensitive disturbances and motor dysfunctions

ELIGIBILITY:
Inclusion Criteria:

* Neck pain

Exclusion Criteria:

* myelopathy
* fracture
* infection
* dystonia
* tumor
* inflammatory disease
* fibromyalgia
* or osteoporosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from Pain intensity at 24 hours | 24 hours, 5 minutes after the treatment
  Pressure Pain Thresholds (PPT) will be assessed bilaterally over the masseter, temporalis, trapezius and suboccipital muscles by an assessor blinded to the subjects condition.
Maximum mouth opening without pain at 24 hours | 24 hours, 5 minutes after the treatment
  Is the ability to open the mouth so widely as you could without pain.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) at 24 hours | 24 hours, 5 minutes after the treatment
  Will be used to measure PCS

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, Principal Investigator — IRCCS Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: Undecided